CLINICAL TRIAL: NCT05219604
Title: The Magnitude and Duration of the Central Nervous System Effects Following Intravenous Infusion of Diphenhydramine Using Pharmacokinetic and Pharmacodynamic Modeling
Brief Title: Central Nervous System Effects Following Infusion of Diphenhydramine Using Pharmacokinetic and Pharmacodynamic Modeling
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Institution decision
Sponsor: Dent Neuroscience Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DIP-PKPD
Record Dates: First submitted 2022-01-18; First posted 2022-02-02 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Effects of Diphenhydramine; Pharmacokinetics of Diphenhydramine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: DiphenhydrAMINE Injectable Solution — Intravenous infusion of diphenhydramine 50 mg.

SUMMARY:
This study seeks to explore the magnitude and duration of central nervous system effects and pharmacokinetics after intravenous infusion of diphenhydramine.

ELIGIBILITY:
Inclusion Criteria:

1. Medically-stable volunteers of either gender between 35 and 50 years old or over the age of 65
2. No medication changes anticipated for the duration of the study except as defined in protocol

Exclusion Criteria:

1. Insulin-dependent diabetes
2. Psychiatric or neurologic disease affecting cognition in a way that may interfere with study outcomes in the opinion of the investigator
3. Unstable Coronary Artery Disease (active angina, MI within 6 months, stent placement within 6 months, cardiac surgery within 6 months)
4. Estimated CrCl < 30 mL/min using the Cockroft-Gault equation based on ideal body weight or total body weight
5. Any malignancy actively being treated or not in remission
6. Currently taking any CNS stimulant or depressant medications that may interfere with study outcomes in the opinion of the investigator unless using as defined in the protocol
7. Positive toxicology test for marijuana at screening visit or visit 2 or using marijuana not as defined in the protocol
8. Active or recent history of a substance use disorder within one year
9. Any medical condition that in the opinion of the investigator would disqualify the subject from participation in the study
10. Female subjects who are pregnant, planning to become pregnant, or breastfeeding on any study day
11. Female subjects of childbearing potential unwilling to use acceptable method of contraception during the study as defined in the protocol
12. Contraindication, known allergy, or suspected intolerability to study medication
13. Receipt of an antihistamine within 5 half-lives prior to the start of study visit 1 or study visit 2, as determined by the investigator
14. Positive toxicology test for a drug that is inconsistent with permitted medication use (defined in the protocol) as interpreted by the investigator
15. Participation in any other investigational drug study during the study or within 4 weeks prior to screening

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Rainka, PharmD, Principal Investigator — Dent Neurologic Institute
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diphenhydramine 50 mg IV Infusion: Participants received an IV infusion containing 50 mg diphenhydramine in NS.
Period: Overall Study
Arm/Group | Diphenhydramine 50 mg IV Infusion
Started | 3
Completed | 3 (Study terminated due to institution decision.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Reaction Time)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  Reaction Time Median Five-Choice Reaction Time is the median duration it took for a subject to release the response button after the presentation of the target stimulus, calculated across correct, assessed trials in which the stimulus could appear in any one of five locations. Lower is better. Minimum score is 100 and maximum score is 5100.
Time Frame: Change from before to after diphenhydramine administration (30, 60, 210, 240, 450, and 480 minutes after diphenhydramine)
Population: Data were collected for 3 study participants prior to study termination. There were no participants with data collected at the following time points due to early study termination as no participants were enrolled in the group to have data collected at these time points: 60 min, 240 min, or 480 min post-diphenhydramine. Data were not analyzed via ANOVA with contrast or via PK/PD modeling as planned as there were lack of sufficient data to perform this analysis due to early study termination.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
ms
  Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time) | 246 (51.4)
  Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 289.7 (87.8)
  Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 267.0 (72.9)
  Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 292.8 (94.6)

2. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Reaction Time)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  Reaction Time Median Five-Choice Reaction Time is the median duration it took for a subject to release the response button after the presentation of the target stimulus, calculated across correct, assessed trials in which the stimulus could appear in any one of five locations. Lower is better. Minimum score is 100 and maximum score is 5100.
Time Frame: Before and after diphenhydramine administration (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
ms
  Elderly Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time) | 264 (58.3)
  Adult Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time) | 211 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 314.0 (108.9)
  Adult Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 241.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 278.3 (99.3)
  Adult Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 244.5 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 321.0 (114.6)
  Adult Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 236.5 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

3. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Digit Span)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  Digit Span Maximum Span Passed Forwards is the longest sequence problem successfully reached and passed by the subject. Higher is better. Minimum score is 0 and maximum score is 9.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (1.4)
  Adult Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.5 (2.1)
  Adult Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 6.0 (1.4)
  Adult Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 7.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 6.0 (1.4)
  Adult Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

4. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Visual Analog Scale for Sedation)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  The Visual Analog Scale for Sedation is a scale where participants indicate their current state on a scale from "Sedated" to "Alert". Higher score is more alert. Minimum score is 0 and maximum score is 12.8.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Visual Analog Scale for Sedation Pre-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation Pre-Diphenhydramine | 12.3 (0.5)
  Adult Visual Analog Scale for Sedation Pre-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation Pre-Diphenhydramine | 12.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine | 2.0 (2.2)
  Adult Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine | 10.8 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine | 6.3 (3.2)
  Adult Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine | 11.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine | 4.8 (6.4)
  Adult Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine | 11.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

5. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Digit Span)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  Digit Span Maximum Span Passed Forwards is the longest sequence problem successfully reached and passed by the subject. Higher is better. Minimum score is 0 and maximum score is 9.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards) | 5 (1.0)
  Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.3 (1.5)
  Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 6.3 (1.2)
  Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.7 (1.2)

6. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Visual Analog Scale for Sedation)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  The Visual Analog Scale for Sedation is a scale where participants indicate their current state on a scale from "Sedated" to "Alert". Higher score is more alert. Minimum score is 0 and maximum score is 12.8.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Visual Analog Scale for Sedation Pre-Diphenhydramine | 12.3 (0.4)
  Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine | 4.9 (5.3)
  Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine | 7.9 (3.7)
  Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine | 6.9 (5.9)

7. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Spatial Working Memory)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  Spatial Working Memory Between Errors is the number of times the subject incorrectly revisits a box in which a token has been previously found. Lower is better. Minimum score is 0 and maximum score is 63.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Spatial Working Memory Pre-Diphenhydramine (Between Errors) | 1.7 (2.9)
  Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors) | 4.0 (6.9)
  Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors) | 1.0 (1.7)
  Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors) | 2.3 (4.0)

8. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Paired Associates Learning)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  Paired Associates Learning First Attempt Memory Score is the number of times a subject chose the correct box on their first attempt when recalling the pattern locations. Higher is better. Minimum score is 0 and maximum score is 20.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score) | 16.0 (3.6)
  Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 11.7 (6.1)
  Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 15.7 (4.0)
  Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 14.0 (4.6)

9. Primary Outcome: Change in Score of Battery of Cognitive Function Tests (Rapid Visual Information Processing)
Description: Change in the results of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation after diphenhydramine administration compared to baseline.
  Rapid Visual Processing Median Response Latency is the median response latency on trials where the subject responded correctly, calculated across all assessed trials. Lower is better. Minimum score is 0 and maximum score is 908.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency) | 482.3 (16.5)
  Rapid Visual Information Processing 30 Minutes Post-Diphenhydramine (Median Response Latency) | 532.2 (50.3)
  Rapid Visual Information Processing 210 Minutes Post-Diphenhydramine (Median Response Latency) | 504.7 (37.5)
  Rapid Visual Information Processing 450 Minutes Post-Diphenhydramine (Median Response Latency) | 471.8 (41.3)

10. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Spatial Working Memory)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  Spatial Working Memory Between Errors is the number of times the subject incorrectly revisits a box in which a token has been previously found. Lower is better. Minimum score is 0 and maximum score is 63.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Spatial Working Memory Pre-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory Pre-Diphenhydramine (Between Errors) | 2.5 (3.5)
  Adult Spatial Working Memory Pre-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory Pre-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors) | 6.0 (8.5)
  Adult Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors) | 0 (0)
  Adult Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors) | 3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors) | 3.5 (4.9)
  Adult Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

11. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Paired Associates Learning)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  Paired Associates Learning First Attempt Memory Score is the number of times a subject chose the correct box on their first attempt when recalling the pattern locations. Higher is better. Minimum score is 0 and maximum score is 20.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score) | 18.0 (1.4)
  Adult Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score) | 12.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 11.0 (8.5)
  Adult Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 13.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 14.5 (4.9)
  Adult Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 18.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 14.5 (6.4)
  Adult Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 13.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

12. Secondary Outcome: Elderly vs. Adult Score of Battery of Cognitive Function Tests at Specified Time Points (Rapid Visual Information Processing)
Description: Score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (0, 30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration).
  Rapid Visual Processing Median Response Latency is the median response latency on trials where the subject responded correctly, calculated across all assessed trials. Lower is better. Minimum score is 0 and maximum score is 908.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency) | 490.5 (12.0)
  Adult Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency) | 466 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency) | 532.3 (71.1)
  Adult Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency) | 532 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency) | 516.0 (45.3)
  Adult Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency) | 482 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency) | 472.8 (58.3)
  Adult Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency) | 470 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

13. Secondary Outcome: Elderly vs. Adult Diphenhydramine AUC
Description: Difference between diphenhydramine pharmacokinetic area under the curve (AUC) in elderly subjects aged 65+ vs. adult subjects aged 35 to 50
Time Frame: Immediately after diphenhydramine administration to 480 minutes after diphenhydramine administration
Population: Blood was collected from study participants as specified in the study protocol; however, samples were destroyed and not analyzed due to early study termination. Therefore, there are no results for this endpoint to report.
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 0

14. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Reaction Time)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  Reaction Time Median Five-Choice Reaction Time is the median duration it took for a subject to release the response button after the presentation of the target stimulus, calculated across correct, assessed trials in which the stimulus could appear in any one of five locations. Lower is better. Minimum score is 100 and maximum score is 5100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
ms
  Elderly Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time) | 264 (58.3)
  Adult Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time Pre-Diphenhydramine (Median Five-Choice Movement Time) | 211 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 314.0 (108.9)
  Adult Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 30 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 241.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 278.3 (99.3)
  Adult Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 210 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 244.5 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 2
  Elderly Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 321.0 (114.6)
  Adult Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time): number analyzed (Participants) | 1
  Adult Reaction Time 450 Minutes Post-Diphenhydramine (Median Five-Choice Movement Time) | 236.5 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

15. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Digit Span)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  Digit Span Maximum Span Passed Forwards is the longest sequence problem successfully reached and passed by the subject. Higher is better. Minimum score is 0 and maximum score is 9.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (1.4)
  Adult Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span Pre-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.5 (2.1)
  Adult Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 30 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 6.0 (1.4)
  Adult Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 210 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 7.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 2
  Elderly Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 6.0 (1.4)
  Adult Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards): number analyzed (Participants) | 1
  Adult Digit Span 450 Minutes Post-Diphenhydramine (Maximum Span Passed Forwards) | 5.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

16. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Visual Analog Scale for Sedation)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  The Visual Analog Scale for Sedation is a scale where participants indicate their current state on a scale from "Sedated" to "Alert". Higher score is more alert. Minimum score is 0 and maximum score is 12.8.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Visual Analog Scale for Sedation Pre-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation Pre-Diphenhydramine | 12.3 (0.5)
  Adult Visual Analog Scale for Sedation Pre-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation Pre-Diphenhydramine | 12.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine | 2.0 (2.2)
  Adult Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 30 Minutes Post-Diphenhydramine | 10.8 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine | 6.3 (3.2)
  Adult Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 210 Minutes Post-Diphenhydramine | 11.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine: number analyzed (Participants) | 2
  Elderly Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine | 4.8 (6.4)
  Adult Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine: number analyzed (Participants) | 1
  Adult Visual Analog Scale for Sedation 450 Minutes Post-Diphenhydramine | 11.3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

17. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Spatial Working Memory)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  Spatial Working Memory Between Errors is the number of times the subject incorrectly revisits a box in which a token has been previously found. Lower is better. Minimum score is 0 and maximum score is 63.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Spatial Working Memory Pre-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory Pre-Diphenhydramine (Between Errors) | 2.5 (3.5)
  Adult Spatial Working Memory Pre-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory Pre-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors) | 6.0 (8.5)
  Adult Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 30 Minutes Post-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors) | 0 (0)
  Adult Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 210 Minutes Post-Diphenhydramine (Between Errors) | 3 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 2
  Elderly Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors) | 3.5 (4.9)
  Adult Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors): number analyzed (Participants) | 1
  Adult Spatial Working Memory 450 Minutes Post-Diphenhydramine (Between Errors) | 0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

18. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Paired Associates Learning)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  Paired Associates Learning First Attempt Memory Score is the number of times a subject chose the correct box on their first attempt when recalling the pattern locations. Higher is better. Minimum score is 0 and maximum score is 20.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score) | 18.0 (1.4)
  Adult Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning Pre-Diphenhydramine (First Attempt Memory Score) | 12.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 11.0 (8.5)
  Adult Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 30 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 13.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 14.5 (4.9)
  Adult Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 210 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 18.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 2
  Elderly Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 14.5 (6.4)
  Adult Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score): number analyzed (Participants) | 1
  Adult Paired Associates Learning 450 Minutes Post-Diphenhydramine (First Attempt Memory Score) | 13.0 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

19. Secondary Outcome: Elderly vs. Adult Change in Score of Battery of Cognitive Function Tests After Diphenhydramine (Rapid Visual Information Processing)
Description: Change in the score of the CANTAB battery of cognitive function tests (reaction time, rapid visual information processing, paired associates learning, spatial working memory, digit span) and visual analog scale for sedation in elderly subjects aged 65+ compared to adult subjects aged 35 to 50 at specified time points (30, 60, 210, 240, 450, 480 minutes after diphenhydramine administration) compared to baseline.
  Rapid Visual Processing Median Response Latency is the median response latency on trials where the subject responded correctly, calculated across all assessed trials. Lower is better. Minimum score is 0 and maximum score is 908.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diphenhydramine 50 mg IV Infusion
Number analyzed (Participants) | 3
units on a scale
  Elderly Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency) | 490.5 (12.0)
  Adult Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing Pre-Diphenhydramine (Median Response Latency) | 466 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency) | 532.3 (71.1)
  Adult Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 30 Min Post-Diphenhydramine (Median Response Latency) | 532 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency) | 516.0 (45.3)
  Adult Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 210 Min Post-Diphenhydramine (Median Response Latency) | 482 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.
  Elderly Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 2
  Elderly Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency) | 472.8 (58.3)
  Adult Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency): number analyzed (Participants) | 1
  Adult Rapid Visual Information Processing 450 Min Post-Diphenhydramine (Median Response Latency) | 470 (NA) — Data from 1 subject are available; therefore, standard deviation is not applicable.

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Diphenhydramine 50 mg IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The study was terminated due to institution decision prior to data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05219604/Prot_SAP_000.pdf